CLINICAL TRIAL: NCT05349292
Title: Effect of Low-volume Fluid Replacement Strategy During Acute Normovolemic Hemodilution on Urine Neutrophil Gelatinase-associated Lipocalin Levels: an Acute Kidney Injury Biomarker
Brief Title: Acute Normovolemic Hemodilution on Urine Neutrophil Gelatinase-associated Lipocalin Levels
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Patrick Odonkor, Associate Professor, University of Maryland, Baltimore
Other Study IDs: HP-00099231
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Acute Normovolemic Hemodilution: Patients undergoing CABG surgery with acute normovolemic hemodilution and autologous blood donation
  Interventions: Other: ANH
- non Acute Normovolemic Hemodilution: Patients undergoing CABG surgery without acute normovolemic hemodilution and autologous blood donation

INTERVENTIONS:
Other: ANH — one group will be managed with ANH and the other without (control group)
  Groups: Acute Normovolemic Hemodilution

SUMMARY:
Acute normovolemic hemodilution (ANH) is performed as a blood conservation technique during surgical procedures with high risk for significant blood loss. It is done by taking out some of the patients blood before surgery actually begins and storing this blood inside of the operating room and giving it back to the patient at the end of surgery when most of the expected surgical bleeding has already occurred. This practice reduces the amount of bleeding that occurs after surgery and also reduces the amount of blood transfusions given to the patient after surgery. Transfusion of blood products from the blood bank may cause problems such as transfusion reactions and infections like hepatitis, and also increases cost.

3 meta-analyses and several smaller trials have shown improvement in blood transfusion rates with the use of ANH, however there is no evidence of improvement in other complication rates, morbidity and mortality, length of stay or cost.

In most types of surgery, when ANH is done, large volumes of IV fluids are given to the patient to prevent a drop in circulatory volume and blood pressure. However during heart surgery, this can cause significant levels of hemodilution in addition to that caused by use of the heart-lung machine. In order to minimize hemodilution when ANH is performed during heart surgery, a smaller amount of IV fluids are given to the patient after blood is drawn. Vasoactive medications are then administered to prevent the blood pressure from dropping.

Kidney injury is a recognized complication that may occur after heart surgery. It may be caused by low blood volume, low blood pressure and anemia. It is not known whether performance of ANH and use of the heart-lung machine may increase risk for kidney injury. Kidney injury is associated with increased risk for other medical complications and death. This increased risk for kidney injury arising from ANH has not been evaluated. This study will therefore compare patients treated with ANH to those not treated with ANH to determine whether there is an increased risk for kidney injury with the use of ANH.

DETAILED DESCRIPTION:
The study population will consist of 50 adult patients less than 70 years old undergoing elective coronary artery bypass graft (CABG) surgery with anticipated CPB duration less than 2 hours at the University of Maryland Medical Center (UMMC). Patients less than 70kg in weight and patients with renal insufficiency and/or hemoglobin levels less than 12g/dL will be excluded. We shall also exclude patients with heart failure (EF <40%) and any significant hepatic or pulmonary comorbidities, including pulmonary hypertension. Patients undergoing emergency and redo cardiac surgery and those with inherited or acquired bleeding disorders will also be excluded.

This study will be a non-blinded randomized prospective observational study. Due to the nature of the intervention being evaluated, blinding will not be achievable. We shall randomly divide patients into 2 groups, where one group will be managed with ANH and the other without (control group). Patients managed with ANH will have 12cc/kg of blood salvaged and stored at room temperature prior to CPB. The stored blood will then be administered to the patient after CPB. Intravascular volume will be replenished in a 1:1 ratio with balanced crystalloid solution during blood salvage. The other group of patients will receive an empiric 7cc/kg bolus of intravenous balanced crystalloid solution prior to CPB. On average, crystalloid infusions are limited to about 500cc prior to CPB to minimize hemodilution of blood.

Patients will otherwise be managed according to normal protocols and pathways used in the perioperative management of CS patients at UMMC.

ELIGIBILITY:
Inclusion Criteria:

* Elective Coronary Artery Bypass Graft Surgery
* Age 18-70 years
* Anticipated Cardiopulmonary Bypass Duration less than 2 hours
* Weight greater than 70kg
* Hemoglobin greater than 12 g/dL

Exclusion Criteria:

* Emergency and redo cardiac surgery
* Renal insufficiency with serum creatinine greater than 1.25 mg/dL and/ or estimated GFR less than 60 mL/min/1.73 m2
* Heart Failure with EF <40%
* Hepatic disease
* Pulmonary Disease, including pulmonary hypertension
* Inherited or Acquired Bleeding Disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 50 adult patients less than 70 years old undergoing elective coronary artery bypass graft (CABG) surgery with anticipated CPB duration less than 2 hours at the University of Maryland Medical Center (UMMC).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Urinary Biomarkers NGAL and KIM-1 | 24 hours
  Urinary levels of NGAL and KIM-1 biomarkers during the first 24 hours after CABG surgery

SECONDARY OUTCOMES:
AKI by KDIGO criteria | 72 hours
  Creatinine values and urine output for 3 days after CS will be recorded for calculation of AKI by KDIGO criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Odonkor, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grant MC, Resar LM, Frank SM. The Efficacy and Utility of Acute Normovolemic Hemodilution. Anesth Analg. 2015 Dec;121(6):1412-4. doi: 10.1213/ANE.0000000000000935. No abstract available. PMID 26579641